CLINICAL TRIAL: NCT04958642
Title: A Phase 2B/3 Prospective, Randomized, Double-Blind, Sham-Controlled Trial of VTS-270 (2-hydroxypropyl-β-cyclodextrin) in Subjects With Neurologic Manifestations of Niemann-Pick Type C1 (NPC1) Disease
Brief Title: Adrabetadex to Treat Niemann-Pick Type C1 (NPC1) Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated by previous Sponsor decision
Sponsor: Mandos LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTS301 (Part C); 2015-002548-15 (EudraCT Number)
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Results first posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Niemann-Pick Disease, Type C
Keywords: Niemann-Pick Type C1 (NPC1) Disease; neurologic disease; gross motor dysfunction; fine motor dysfunction; dysphagia; swallowing problems; cognitive dysfunction; gait abnormalities; pediatrics
MeSH Terms: conditions — Niemann-Pick Disease, Type C; Disease; Deglutition Disorders; Cognitive Dysfunction; Mobility Limitation | interventions — 2-Hydroxypropyl-beta-cyclodextrin; Cyclodextrins

STUDY DESIGN:
Intervention Model Description: In Part C, all participants receive adrabetadex
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adrabetadex (Experimental): All participants receive their prescribed dose of adrabetadex. Dose is allowed to be adjusted down to a minimum of 400 milligrams (mg) or up to a maximum of 900 mg, at the investigator's discretion.
  Interventions: Drug: Adrabetadex

INTERVENTIONS:
Drug: Adrabetadex — Mallinckrodt test formulation, administered intrathecal (IT) via lumbar puncture (LP) infusion.
  Other Names: VTS-270; 2-hydroxypropyl-β-cyclodextrin; Cyclodextrin

SUMMARY:
Due to different study designs, the sponsor separated Part C into this separate registration (NCT04958642), leaving Parts A/B in NCT02534844. The trial's final results for the primary outcome measure of Adverse Events (AE) will be reported here.

This study is to evaluate how safe and effective adrabetadex is for participants with Niemann-Pick Type C1 (NPC1) disease who experience neurologic symptoms (listed under Keywords).

In Parts A/B (NCT02534844), two out of every 3 participants will receive the study drug. The third participant will receive 1 to 2 small needle pricks at the location where the IT injection is normally made (sham control).

In Part C, all participants will receive study drug.

DETAILED DESCRIPTION:
Participants in Part C will receive adrabetadex until the investigator considers adrabetadex to no longer be beneficial to the participant, or the development program is discontinued.

ELIGIBILITY:
Inclusion criteria:

One of the following is required for inclusion into VTS301 Part C:

* Has agreed to convert from the monthly dosing regimen used in the NIH phase 1/2a protocol to an every 2 weeks dosing regimen
* The investigator has received prior written authorization from the sponsor for the participant to enter VTS301 Part C on an amended dose and/or regimen
* Has received prior written authorization from Vtesse to enroll directly into Part C

Exclusion criteria:

* None of the inclusion criteria are applicable

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Lead, Study Director — Mandos LLC
Locations (30):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Orange County: CHOC Children's, Orange, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands Children's Hospital, Gainesville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Eunice Kennedy Shriver National Institute of Child Health and Human Development, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Multicare Institute for Research and Innovation, Tacoma, Washington
- Australia (4):
  - The Prince of Wales Hospital, Randwick, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Melbourne, Victria
  - Royal Perth Hospital, Perth, Western Australia
- CHU Paris Est - Hopital d'Enfants Armand-Trousseau, Paris, Cedex 12, France
- Germany (3):
  - Katholisches Klinikim Bochum gGmbH, Bochum
  - Universitaetsklinikum Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
- Waikato Hospital, Hamilton, New Zealand
- National University Hospital (Singapore) Pte, Ltd, Singapore, Singapore
- INSELSPITAL, Universitätsspital Bern, Bern, Switzerland
- Turkey (Türkiye) (2):
  - Gazi University Medical Faculty, Ankara
  - Hacettepe University Medical Faculty, Ankara
- United Kingdom (2):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Great Ormond Street Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is an open-label extension phase of study VTS301 (Parts A/B) (NCT02534844). Participants who completed Part B and participants who completed National Institutes of Health (NIH) phase 1 study (Protocol 13-CH-0001) were eligible to participate in this study.
Groups:
- Treatment Naive: Treatment-naive participants received adrabetadex 900 milligrams (mg) administered intrathecal (IT) via lumbar puncture (LP) infusion every 2 weeks until the investigator considered adrabetadex to no longer be beneficial to the participant, or the development program was discontinued.
- Previously Treated in Phase I: Rollover participants from Study 13-CH-0001 received adrabetadex at an amended dose and/or regimen after prior written authorization from the sponsor. The treatment was continued until the investigator considered adrabetadex to no longer be beneficial to the participant, or the development program was discontinued.
- Previously Treated in Part A/B: Participants continuing from Part B of the study received adrabetadex 900 mg administered IT via LP infusion every 2 weeks until the investigator considered adrabetadex to no longer be beneficial to the participant, or the development program was discontinued.
Period: Overall Study
Arm/Group | Treatment Naive | Previously Treated in Phase I | Previously Treated in Part A/B
Started | 18 | 13 | 35
Received at Least 1 Dose of Study Drug | 18 | 13 | 35
Completed | 0 | 0 | 0
Not Completed | 18 | 13 | 35
Not completed — Transferred to OLEX program | 3 | 0 | 5
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 9 | 13
Not completed — Investigator's Decision | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Termination by Sponsor/Regulatory Authorities | 8 | 4 | 13
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Transferred to EAP following study termination | 0 | 0 | 1
Not completed — Transferred to Expanded Access Program | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Open-label population included participants who received at least 1 dose of adrabetadex during Part C.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Naive | Previously Treated in Phase I | Previously Treated in Part A/B | Total
Number analyzed (Participants) | 18 | 13 | 35 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (5.07) | 17.5 (6.16) | 14.1 (5.60) | 14.5 (5.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 15 | 32
  Male | 8 | 6 | 20 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 6
  Not Hispanic or Latino | 15 | 11 | 29 | 55
  Unknown or Not Reported | 0 | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 16 | 13 | 29 | 58
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A TEAE was defined as an AE with onset on or after the start of adrabetadex treatment. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to 5 years
Population: The Open-label population included participants who received at least 1 dose of adrabetadex during Part C.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Naive | Previously Treated in Phase I | Previously Treated in Part A/B
Number analyzed (Participants) | 18 | 13 | 35
Participants
  Any TEAEs | 18 | 13 | 34
  SAEs | 9 | 7 | 20

ADVERSE EVENTS:
Time Frame: Baseline up to 5 years
Description: The Open-label population included participants who received at least 1 dose of adrabetadex during Part C.
Arm/Group | Treatment Naive | Previously Treated in Phase I | Previously Treated in Part A/B
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/13 | 1/35
Serious Adverse Events (participants affected / at risk) | 9/18 | 7/13 | 20/35
Other Adverse Events (participants affected / at risk) | 18/18 | 13/13 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Naive (N=18) | Previously Treated in Phase I (N=13) | Previously Treated in Part A/B (N=35)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Superior mesenteric artery syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Herpes simplex pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (5) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stoma site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Intentional medical device removal by patient (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chorea (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Seizure cluster (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal subdural haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 2 (2)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Naive (N=18) | Previously Treated in Phase I (N=13) | Previously Treated in Part A/B (N=35)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 3 (3) | 2 (3)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 3 (3)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 9 (20) | 4 (7) | 9 (12)
Neurosensory hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 6 (72) | 2 (5) | 5 (5)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1) | 2 (2)
Anal incontinence (Gastrointestinal disorders) | 2 (5) | 2 (10) | 2 (6)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 9 (15)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (19) | 6 (14) | 14 (28)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 6 (6) | 6 (10)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Malpositioned teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 4 (13) | 6 (10)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retained deciduous tooth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (26) | 9 (24) | 16 (25)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 1 (1)
Application site rash (General disorders) | 0 (0) | 1 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 2 (2)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 8 (101) | 5 (11) | 13 (146)
Gait disturbance (General disorders) | 2 (4) | 6 (10) | 10 (55)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (3) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (3) | 0 (0)
Pain (General disorders) | 1 (2) | 2 (3) | 3 (4)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (13) | 9 (48) | 17 (36)
Swelling (General disorders) | 1 (2) | 0 (0) | 2 (4)
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 2 (3)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 3 (8)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 3 (4) | 2 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 3 (5) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (10) | 3 (6) | 7 (13)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (2) | 3 (6) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (3) | 4 (4) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 3 (4) | 0 (0) | 7 (7)
Sinusitis (Infections and infestations) | 0 (0) | 3 (4) | 2 (3)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 11 (34) | 7 (27) | 10 (24)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Administration related reaction (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (10) | 7 (17) | 5 (29)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (3) | 2 (2)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (37) | 7 (42) | 16 (117)
Foot fracture (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 5 (10)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 5 (5)
Lip injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Oral contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 3 (33)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (10)
Procedural pain (Injury, poisoning and procedural complications) | 3 (6) | 1 (1) | 5 (15)
Sedation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (9) | 6 (15) | 11 (33)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 4 (7)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 2 (2)
Body temperature increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Electroencephalogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Mean cell volume decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (2) | 1 (1)
PO2 decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1)
Respiratory rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 3 (4) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Polydipsia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (36) | 9 (74) | 18 (142)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (14) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (16) | 2 (5)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (18) | 3 (10) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (7) | 7 (12)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 9 (21) | 2 (7) | 8 (78)
Atonic seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 2 (3) | 8 (15)
Cataplexy (Nervous system disorders) | 3 (3) | 1 (1) | 5 (7)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Diplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (2) | 2 (4)
Dysarthria (Nervous system disorders) | 3 (18) | 1 (3) | 2 (64)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 2 (2) | 4 (5) | 2 (3)
Epilepsy (Nervous system disorders) | 2 (5) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 9 (29) | 9 (34) | 12 (79)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 3 (3) | 1 (4) | 4 (11)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 2 (4)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Movement disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Repetitive speech (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (3) | 4 (34) | 8 (14)
Seizure cluster (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 2 (4)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Communication disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Daydreaming (Psychiatric disorders) | 1 (5) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dyssomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Inappropriate affect (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 2 (3)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (9) | 2 (4)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (2) | 1 (1)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Perineal rash (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic respiratory symptom (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Apnoea (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (4)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (13) | 6 (15) | 15 (29)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4) | 9 (45)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 3 (3) | 6 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2)
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 1 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 3 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin striae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 3 (4)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The development program for adrabetadex was discontinued and Part C of the study was terminated by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT04958642/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT04958642/SAP_001.pdf